CLINICAL TRIAL: NCT00004316
Title: Phase I/II Randomized, Placebo-Controlled Study of Capsaicin for Interstitial Cystitis and Vulvar Vestibulitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 199/11835; R01DK049524 (NIH)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2008-09

CONDITIONS: Interstitial Cystitis; Vulvar Diseases
Keywords: interstitial cystitis; rare disease; renal and genitourinary disorders; vulvar vestibulitis
MeSH Terms: conditions — Cystitis, Interstitial; Vulvar Diseases; Rare Diseases; Urogenital Diseases; Vulvar Vestibulitis | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Capsaicin (Experimental)
  Interventions: Drug: capsaicin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: capsaicin
  Arms: Capsaicin
Drug: Placebo
  Arms: Placebo

SUMMARY:
OBJECTIVES: I. Estimate the optimal safe dose of intravesical capsaicin in patients with interstitial cystitis.

II. Evaluate the efficacy of 0.025% topical capsaicin in relieving chronic burning pain in patients with vulvar vestibulitis.

III. Evaluate the effect of capsaicin on type C nerve fibers in bladder mucosa and vulvar skin.

IV. Evaluate the effect of C fiber depletion on urinary levels of histamine and prostaglandin.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients with interstitial cystitis are randomly assigned to 1 of 3 pain control therapies.

The first group is treated with capsaicin. A second group is given individually titrated doses of capsaicin: the dose is increased as tolerated or until symptomatic response is acceptable. A control group receives a placebo. Therapy for all groups is administered intravesically every week for 5 weeks.

Patients with vulvar vestibulitis are randomly assigned to 1 of 2 pain control therapies. One group applies topical capsaicin cream to the painful area 4 times a day for 6 weeks. The dose is individually titrated if burning discomfort persists and the patient is compliant with the application schedule. The control group applies a placebo.

Patients with vulvar vestibulitis may continue or cross to capsaicin for 6 additional weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Women with interstitial cystitis by National Institute of Diabetes and Digestive and Kidney Diseases criteria Vulvar vestibulitis by International Society for the Study of Vulvar Disease, i.e.: Severe pain on touch or attempted entry of vagina Tenderness to pressure within the vulvar vestibule Vulvar erythema Duration of symptoms at least 6 months Absence of vulvovaginal infection, i.e.: No fungus No trichomonas No chlamydia No gonorrhea No "clue cells" in vaginal discharge

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 1995-06 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Flood, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittspurgh, Pittsburgh, Pennsylvania, United States